CLINICAL TRIAL: NCT03847298
Title: Evaluation of Physical Fitness and Physical Activity Levels of Pediatric Arrhythmia Patients With Pacemaker
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sena Teber, Research Assistant, Hacettepe University
Other Study IDs: GO 17/880
Record Dates: First submitted 2019-01-04; First posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Pacemaker; Physical Activity
Keywords: pediatric; pacemaker; physical activity; physical fitness
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pacemaker
  Interventions: Other: Physical activity and physical fitness assessment
- Control
  Interventions: Other: Physical activity and physical fitness assessment

INTERVENTIONS:
Other: Physical activity and physical fitness assessment — Physical fitness was assessed using Munich Physical Fitness Test (MFT). The SenseWear Armband metabolic holter device was used to record the physical activity level for consecutive 7 days. The functional exercise capacity of the individuals was assessed by the six-minute walking test (6MWT) and cardiorespiratory capacity was assessed by maximal exercise test on the treadmill.

SUMMARY:
The aim of this study was to evaluate physical fitness and physical activity levels of pediatric arrhythmia patients with pacemaker compared with their healthy peers.

DETAILED DESCRIPTION:
Studies in children with heart diseases suggest that physical activity levels are reduced relative to their peers, which in turn increases cardiovascular risk factors and cardiac rhythm problems. To the best of our knowledge, physical fitness and objectively measured physical activity levels of children with a pacemaker have not been studied. The aim of this study was to evaluate physical fitness and physical activity levels of pediatric arrhythmia patients with a pacemaker compared with their healthy peers.

Investigators enrolled clinically stable pediatric patients and used the echocardiogram to evaluate cardiac functions of all patients. Physical fitness was assessed using the Munich Physical Fitness Test (MFT). The SenseWear Armband metabolic Holter device was used to record the physical activity level for consecutive 7 days.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria of the Pacemaker Group:

* Permanent pacemaker
* Being 7-18 years of age
* Able and willing to complete the informed consent process
* Able to walk and co-operate

Exclusion Criteria:

Exclusion criteria of Pacemaker Group:

* Unstable medical condition
* To have severe neurological, severe orthopedic problems
* To have severe heart failure and another systemic disease or acute infection
* Down Syndrome
* The control group will consist of healthy subjects.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with pacemakers who were followed routinely in Hacettepe Hospital, Department of Pediatric Cardiology.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2017-11-19 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-06-24 (Actual)

PRIMARY OUTCOMES:
Physical Activity Level | seven days
  Physical activity index will be measured using activity monitor for seven consecutive days.
Total Number of Steps | seven days
  Participants will wear an accelerometer (physical activity monitor) for seven consecutive days.
Munich Physical Fitness Test Score | 1st day (before using device)
  The test consists of six different parameters, including balancing and bouncing (speed and coordination), accurate throw (speed and coordination), trunk flexibility, vertical jumping (power), hanging (endurance and strength), and step test (endurance, speed and coordination). After all the parameters are completed, the score of each parameter is calculated from the standardization chart according to age and sex. This total score is divided by the number of parameters and recorded as Munich total score. Physical fitness is classified according to scores as deficient (<35), normal (36-45), satisfactory (46-55), good (56-65) and very good (>66).

SECONDARY OUTCOMES:
Functional exercise capacity (6 minutes walk test) | 1st day (before using device)
  6-minute walk test will be performed in a long, straight, enclosed corridor 30 meters in length. Patients are required to walk in their walking speed with standardized instructions. The distance walked by subjects during 6 minutes will be recorded.
Cardiorespiratory Capacity (maximal exercise test on the treadmill) | 8th day (last day of the assessment)
  The symptom limited maximal exercise test will be performed without gas exchange measurement. The Modified Bruce Protocol will be applied on the treadmill.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Unit and Hacettepe University Faculty of Medicine, Department of Pediatrics, Department of Pediatric Cardiology, Ankara, Turkey (Türkiye)